CLINICAL TRIAL: NCT05395325
Title: The Clinical Effects of Combined Kinesiotaping and Steroid Injection in Stroke Patients With Hemiplegic Shoulder Pain : A Randomized Controlled Trial
Brief Title: Clinical Effects of Combined Kinesiotaping and Steroid Injection in Stroke Patients With Hemiplegic Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG8M0431
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Hemiplegic Shoulder Pain
Keywords: hemiplegic shoulder pain; Kinesiotaping; Stroke; steroid injection
MeSH Terms: conditions — Stroke | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT and steroid injection group (Experimental): the patients will receive steroid injection for only one time before intervention, and receive KT for 5 days a week, for three weeks. And a 30-minute hand functional training would also be provided once daily every day during the intervention.
  Interventions: Other: Kinesiotaping; Other: Hand rehabilitation program; Other: Steroid injection
- KT group (Sham Comparator): the patients will receive KT for 5 days a week, for three weeks. And a 30-minute hand functional training would also be provided once daily every day during the intervention.
  Interventions: Other: Kinesiotaping; Other: Hand rehabilitation program

INTERVENTIONS:
Other: Kinesiotaping — Kinesio tape would be applied (1)over the extensor muscles of the affected hand for facilitating the extension of hand. We will apply the tape from the upper 1/3 length of dorsal side of the forearm and split the tape into five equal bars to the distal interphalangeal joint of each finger along the finger bones. (2) from above the scapula spine to the medial deltoid. (3) from medial border of scapula to anterior deltoid.This intervention would be executed for five days per week for three weeks.
Other: Hand rehabilitation program — In the thirty-minute hand rehabilitation program, a motor-relearning theory would be implemented into the intervention by teaching the participants how to use their upper limb properly without any compensatory motions. Therefore, for establishing a correct movement pattern, an occupational therapist would provide a hand-guided activity, in which the participants could practice reaching movement as well as hand grasp and release in a more natural way. Besides, the therapist would also help the patients release their muscle tone by stretching the spastic muscles for five minutes before and after this hand rehabilitation period
Other: Steroid injection — all the steroid injection would be executed by physicians. The 23G needles would be used for the injections. The examiners would be clear and familiar with the protocol, and the injections would be executed for only one time during the study period in experimental group.
  Arms: KT and steroid injection group

SUMMARY:
The aims of this study is to investigate sono-guided shoulder steroid injection combined with Kinesiotaping applications in reducing shoulder pain, improving functional performance on upper extremity and quality of life in stroke patients with hemiplegic shoulder pain.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is one of the most common complications in stroke patients, and it has negative effects on rehabilitation in hemiplegic side, functional recovery of upper extremity, and quality of life. The common treatments for hemiplegic shoulder pain include oral medication,transcutaneous electrical nerve stimulation, and local injections. Steroid or sodium hyaluronate are mainly used in local injections. Steroid can suppress inflammation and immune system effectively.

Furthermore, the clinical characteristics of impaired motor performance on affected limb in stroke patients include muscle weakness, increased muscle tone, contracture, joint instability, or impaired of motor control. Impaired motor performance of upper extremity and spasticity have negative impacts in functional performances and daily activities. In stroke patients with poststroke spasticity, stretching, range of motion exercises, antispasticity splint, neuromuscular electrical stimulation, oral medications and local injection of botulinum toxin are recommended. Some investigators found that Kinesiotaping (KT) combined with other interventions may facilitate muscle function, provide joint support and proprioception feedback, and reduce pain in stroke patients with hemiplegia. Thus, the investigators will perform steroid injection in stroke patients with hemiplegic shoulder pain to reduce pain, and apply KT while receiving rehabilitation to facilitate motor recovery and functional performance in affected upper extremity.

In this study, 50 stroke patients with hemiplegic shoulder pain will be recruited and randomly divided into experimental and control groups. In experimental group(n=25), the patients will receive KT combined steroid injection with rehabilitation, and the injection will perform only one time in the entire intervention period. In control group, the patients will receive KT with rehabilitation. In both groups, KT will be applied for three weeks. All participants will receive shoulder sonography evaluation before intervention to investigate the condition of hemiplegic shoulder pain and receive physical examination, hand function assessment before intervention, after the three-week intervention and three-week post intervention.

The aims of this study is to investigate sono-guided shoulder steroid injection combined with Kinesiotaping applications in reducing shoulder pain, improving functional performance on upper extremity and quality of life in stroke patients with hemiplegic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* The patients have a stroke with hemiplegia (duration is less than 6 months after stroke).
* The patients complain about shoulder pain and there're soft tissue impairment under sonography measurement.
* Patients who are able to perform slightly hand grasp( at least 10 degrees at metacarpophalangeal and interphalangeal joints).

Exclusion Criteria:

* age is younger than 20 years old or older than 80 years old
* previous history of upper extremity tendon or neuromuscular injury, shoulder pain, frozen shoulder or shoulder surgery before stroke,
* any other systemic neuromuscular disease; cognition or language impairment leading to communication difficulty.
* allergic to kinesio tape

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
the change from baseline to time of Fugl-Meyer assessment for upper extremity | 4th week, and 7th week
  a therapist will evaluate Fugl-Meyer assessment for upper extremity (FMA-UE) for each participant. In this assessment, participants would need to execute a series of movements, which involved proximal and distal part of upper limb. The higher the grade, the better the performance. The total score ranges from 0 to 66 for motor function.
the change from baseline to time of Flexilevel Scale of Shoulder Function | 4th week, and 7th week
  Flexilevel Scale of Shoulder Function(FLEX-SF) would be used to measure the shoulder performance in daily activities.It is a self-reported questionnaire. The higher the grade, the better the performance.

SECONDARY OUTCOMES:
the change from baseline to time of Brunnstrom stage | 4th week, and 7th week
  a therapist will measure motor recovery stage (Brunnstrom stage)
the change from baseline to time of quality of life by Stroke Impact Scale | 4th week, and 7th week
  Stroke Impact Scale would be used to measure the independence of daily activities. It is a self-reported questionnaire. The contents involve various aspect of life. The high the grade, the more serious the life is affected. The total score is from 0 to 100 for self-assessing the level of recovery.
the change from baseline to time of quality of life by Barthel Index | 4th week, and 7th week
  Barthel Index would be used to measure the independence of daily activities. It is a form that contains different activities of daily living. The higher the outcome grades, the better the level of independence.
the change from baseline to time of functional performance by box and block test | 4th week, and 7th week
  box and block test would be used to assess the grasping and release performance of the affected hand.
the change from baseline to time of functional performance by STEF | 4th week, and 7th week
  Simple Test for Evaluating Hand Function (STEF) would be used to assess the hand function by executing various types of grasping.
the change from baseline to time of VAS | 4th week, and 7th week
  Visual Analog Scale (VAS) would be used to assess the self-reported shoulder pain level of patients. The score ranges from 0 to 10. The higher the grades, the worst pain the patients experienced.
the change from baseline to time of PROM | 4th week, and 7th week
  a therapist will measure passive range of motions of shoulder joint.
the change from baseline to time of edema | 4th week, and 7th week
  a therapist will measure forearm, wrist and middle palm circumference to assess edema.
the change from baseline to time of MAS scale | 4th week, and 7th week
  a therapist will measure spasticity of affected upper extremity at elbow and wrist joints (modified Ashworth scale). In this scale, muscle tone would be assessed by quick stretch of muscle belly. The scoring criteria are as follows. 0, no increase in muscle tone; 1, Slight increase in muscle tone; 2, More marked increase in muscle tone through most of the ROM; 3, considerable increase in muscle tone; 4, affected part(s) rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Huang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No